CLINICAL TRIAL: NCT04235959
Title: A Multiple Dose Titration Study in Chinese Patients With Type 2 Diabetes Mellitus to Investigate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Efficacy of Tirzepatide
Brief Title: A Study of Tirzepatide in Chinese Participants With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 17379; I8F-MC-GPHT (Other: Eli Lilly and Company)
Record Dates: First submitted 2020-01-20; First posted 2020-01-22 (Actual); Results first posted 2023-07-06 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2022-08

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Tirzepatide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo (Placebo Comparator): Participants received placebo once weekly (QW) subcutaneously (SC).
  Interventions: Drug: Placebo
- Tirzepatide - Cohort 1 (2.5 to 10 Milligram (mg)) and Cohort 2 (2.5 to 15 mg) (Experimental): Participants in Cohort 1 received weekly SC doses of tirzepatide with titration regimen starting from 2.5 mg for Weeks 0 through 3 followed by 5 mg for Weeks 4 through 7, 7.5 mg for Weeks 8 through 11, and 10 mg for Weeks 12 through 15.
  Participants in Cohort 2 received weekly SC doses of tirzepatide with titration regimen starting from 2.5 mg for Weeks 0 through 3 followed by 5 mg for Weeks 4 through 7, 7.5 mg for Weeks 8 through 11, and 10 mg for Weeks 12 through 15, 12.5 mg for Weeks 16 through 19, and 15 mg for Weeks 20 through 23.
  Interventions: Drug: Tirzepatide

INTERVENTIONS:
Drug: Tirzepatide — Administered SC
  Other Names: LY3298176
  Arms: Tirzepatide - Cohort 1 (2.5 to 10 Milligram (mg)) and Cohort 2 (2.5 to 15 mg)
Drug: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
The main purpose of this study is to learn more about the safety and side effects of tirzepatide in Chinese participants with type 2 diabetes mellitus. The study will also measure how much tirzepatide gets into the bloodstream and how long it takes the body to remove it. The study will last about six or eight months for each participant.

ELIGIBILITY:
Inclusion Criteria:

* Have type 2 diabetes mellitus (T2DM) controlled with diet and exercise alone or are stable on a single oral antihyperglycemic medication (OAM), metformin, acarbose, or sulphonylureas only (other types of OAM [dipeptidyl peptidase IV inhibitors, sodium-glucose cotransporter-2 inhibitors, and thiazolidinediones] are not allowed in this study), for at least 3 months
* Have a body mass greater than or equal to (≥)23 kilograms per square meter (kg/m²), inclusive

Exclusion Criteria:

* Have type 1 diabetes mellitus
* Have a history of severe hypoglycemia and/or hypoglycemia unawareness within the 6 months prior to Visit 1
* Have a history of heart block or PR interval greater than (>)220 milliseconds (msec) or any abnormality in the 12-lead electrocardiogram (ECG) at screening that, in the opinion of the investigator, increases the risks associated with participating in the study
* Have a history or presence of pancreatitis or gastrointestinal (GI) disorder or a GI disease that impacts gastric emptying or could be aggravated by glucagon-like peptide-1 (GLP-1) analogs or dipeptidyl peptidase IV (DPP-IV) inhibitors
* Have known allergies to tirzepatide, GLP-1 analogs, or related compounds or any components of the formulation

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-10-21 (Actual); Primary Completion 2021-08-17 (Actual); Study Completion 2021-08-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- China (2):
  - West China Hospital Sichuan University, Chengdu, Sichuan
  - Peking University First Hospital, Beijing

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Feng P, Sheng X, Ji Y, Urva S, Wang F, Miller S, Qian C, An Z, Cui Y. A Phase 1 Multiple Dose Study of Tirzepatide in Chinese Patients with Type 2 Diabetes. Adv Ther. 2023 Aug;40(8):3434-3445. doi: 10.1007/s12325-023-02536-8. Epub 2023 Jun 7. PMID 37285081

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1 (2.5 to 10 Milligram (mg) Tirzepatide): Participants in Cohort 1 received weekly SC doses of tirzepatide with titration regimen starting from 2.5 mg for Weeks 0 through 3 followed by 5 mg for Weeks 4 through 7, 7.5 mg for Weeks 8 through 11, and 10 mg for Weeks 12 through 15.
- Cohort 2 (2.5 to 15 mg Tirzepatide): Participants in Cohort 2 received weekly SC doses of tirzepatide with titration regimen starting from 2.5 mg for Weeks 0 through 3 followed by 5 mg for Weeks 4 through 7, 7.5 mg for Weeks 8 through 11, 10 mg for Weeks 12 through 15, 12.5 mg for Weeks 16 through 19, and 15 mg for Weeks 20 through 23.
Period: Overall Study
Arm/Group | Placebo | Cohort 1 (2.5 to 10 Milligram (mg) Tirzepatide) | Cohort 2 (2.5 to 15 mg Tirzepatide)
Started | 4 | 10 | 10
Received At Least One Dose of Study Drug | 4 | 10 | 10
Completed | 3 | 9 | 10
Not Completed | 1 | 1 | 0
Not completed — Protocol Violation | 0 | 1 | 0
Not completed — Adverse Event | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Groups:
- Placebo: Participants received placebo QW SC.
- Total: Total of all reporting groups
Arm/Group | Placebo | Cohort 1 (2.5 to 10 Milligram (mg) Tirzepatide) | Cohort 2 (2.5 to 15 mg Tirzepatide) | Total
Number analyzed (Participants) | 4 | 10 | 10 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.5 (7.5) | 55.8 (5.2) | 56.8 (5.4) | 56.3 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 6 | 4 | 11
  Male | 3 | 4 | 6 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 10 | 10 | 24
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 4 | 10 | 10 | 24
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  China | 4 | 10 | 10 | 24

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration.
Description: The number of participants with one or more SAEs is assessed as related to the study drug and is summarized cumulatively. A serious adverse event is defined as an event that results in death, initial or prolonged hospitalization, is life-threatening, leads to persistent or significant disability/incapacity, is associated with congenital anomaly/birth defect, or is considered significant by the investigator for any other reason. A summary of SAEs and other non-serious adverse events (AEs), regardless of causality, is reported in the Reported Adverse Events module.
Time Frame: Baseline up to 43 Weeks
Population: All participants who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Placebo | Cohort 1 (2.5 to 10 Milligram (mg) Tirzepatide) | Cohort 2 (2.5 to 15 mg Tirzepatide)
Number analyzed (Participants) | 4 | 10 | 10
participants | 1 | 0 | 0

2. Secondary Outcome: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve From Time Zero to 168 Hour Post-dose (AUC [0-168]) of Tirzepatide (Cohort 1)
Description: PK: AUC [0-168] of Tirzepatide.
Time Frame: Week 0 - (Pre-dose, 8, 24, 48, 72, 168 hours post-dose); Week 7 - (Pre-dose, 8, 24, 48, 72, 168 hours post-dose); Week 15 - (Pre-dose, 8, 24, 48, 72, 168 hours post-dose).
Population: All participants who received at least one dose of tirzepatide and had evaluable PK data in Cohort 1.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram hour per milliliter (ng*h/mL)
Groups:
- Cohort 1: 2.5 to 10 mg Tirzepatide: Participants in Cohort 1 received weekly SC doses of tirzepatide with titration regimen starting from 2.5 mg for Weeks 0 through 3 followed by 5 mg for Weeks 4 through 7, 7.5 mg for Weeks 8 through 11, and 10 mg for Weeks 12 through 15.
Arm/Group | Cohort 1: 2.5 to 10 mg Tirzepatide
Number analyzed (Participants) | 10
nanogram hour per milliliter (ng*h/mL)
  Week 0 | 35100 (14)
  Week 7: number analyzed (Participants) | 9
  Week 7 | 125000 (16)
  Week 15: number analyzed (Participants) | 9
  Week 15 | 263000 (17)

3. Secondary Outcome: PK: AUC [0-168] of Tirzepatide (Cohort 2)
Description: PK: AUC [0-168] of Tirzepatide.
Time Frame: Week 0 - (Pre-dose, 8, 24, 48, 72, 168 hours post-dose); Week 7 - (Pre-dose, 8, 24, 48, 72, 168 hours post-dose); Week 23 - (Pre-dose, 8, 24, 48, 72, 168 hours post-dose).
Population: All participants who received at least one dose of tirzepatide and had evaluable PK data in Cohort 2.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram hour per milliliter (ng*h/mL)
Groups:
- Cohort 2: 2.5 to 15 mg Tirzepatide: Participants in Cohort 2 received weekly SC doses of tirzepatide with titration regimen starting from 2.5 mg for Weeks 0 through 3 followed by 5 mg for Weeks 4 through 7, 7.5 mg for Weeks 8 through 11, 10 mg for Weeks 12 through 15, 12.5 mg for Weeks 16 through 19, and 15 mg for Weeks 20 through 23.
Arm/Group | Cohort 2: 2.5 to 15 mg Tirzepatide
Number analyzed (Participants) | 10
nanogram hour per milliliter (ng*h/mL)
  Week 0 | 30900 (14)
  Week 7 | 110000 (16)
  Week 23 | 357000 (16)

4. Secondary Outcome: PK: Maximum Concentration (Cmax) of Tirzepatide (Cohort 1)
Description: PK: Cmax of Tirzepatide.
Time Frame: as for outcome 2
Population: All participants who received at least one dose of tirzepatide and had evaluable PK data in Cohort 1.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Cohort 1: 2.5 to 10 mg Tirzepatide
Number analyzed (Participants) | 10
nanograms per milliliter (ng/mL)
  Week 0 | 306 (28)
  Week 7: number analyzed (Participants) | 9
  Week 7 | 1030 (13)
  Week 15: number analyzed (Participants) | 9
  Week 15 | 2200 (16)

5. Secondary Outcome: PK: Cmax of Tirzepatide (Cohort 2)
Description: PK: Cmax of Tirzepatide.
Time Frame: as for outcome 3
Population: All participants who received at least one dose of tirzepatide and had evaluable PK data in Cohort 2.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Cohort 2: 2.5 to 15 mg Tirzepatide
Number analyzed (Participants) | 10
nanograms per milliliter (ng/mL)
  Week 0 | 257 (17)
  Week 7 | 915 (18)
  Week 23 | 2930 (20)

ADVERSE EVENTS:
Time Frame: Up To 43 Weeks
Description: All participants who received at least one dose of study drug. Per protocol, Adverse Event analysis was planned as per treatment regimen received.
Arm/Group | Placebo | Cohort 1 (2.5 to 10 Milligram (mg) Tirzepatide) | Cohort 2 (2.5 to 15 mg Tirzepatide)
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 1/4 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 4/4 | 10/10 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=4) | Cohort 1 (2.5 to 10 Milligram (mg) Tirzepatide) (N=10) | Cohort 2 (2.5 to 15 mg Tirzepatide) (N=10)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=4) | Cohort 1 (2.5 to 10 Milligram (mg) Tirzepatide) (N=10) | Cohort 2 (2.5 to 15 mg Tirzepatide) (N=10)
Bundle branch block left (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 2 (2) | 5 (6)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 6 (17) | 4 (5)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 4 (4)
Regurgitation (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Tooth loss (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 1 (2)
Fatigue (General disorders) | 0 (0) | 2 (2) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 2 (2)
Liver injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Amylase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Electrocardiogram qt prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram t wave abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 1 (1) | 3 (5)
Occult blood positive (Investigations) | 0 (0) | 1 (1) | 0 (0)
White blood cells urine positive (Investigations) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 5 (7) | 8 (9)
Hyperlipidaemia (Metabolism and nutrition disorders) | 3 (5) | 5 (6) | 2 (3)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Poor quality sleep (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2020-07-01): https://cdn.clinicaltrials.gov/large-docs/59/NCT04235959/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-30): https://cdn.clinicaltrials.gov/large-docs/59/NCT04235959/SAP_001.pdf